CLINICAL TRIAL: NCT04955574
Title: Probiotic and Antibiotic Therapies in Women With Unexplained Infertility
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Change in departmental research focus.
Sponsor: McMaster University (Other)
Collaborators: One Fertility (Other)
Responsible Party: Principal Investigator, Jocelyn Wessels, Postdoctoral Fellow, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JW-001
Record Dates: First submitted 2021-06-11; First posted 2021-07-09 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Unexplained Infertility; Endometriosis
Keywords: Uterine microbiota; Endometrial microbiota
MeSH Terms: conditions — Endometriosis | interventions — Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Probiotic + Antibiotic Placebo (Experimental)
  Interventions: Other: SH-DS01 + Antibiotic Placebo
- Probiotic + Antibiotic (Experimental)
  Interventions: Drug: SH-DS01 + Metronidazole
- Probiotic Placebo + Antibiotic Placebo (Placebo Comparator)
  Interventions: Other: Probiotic Placebo + Antibiotic Placebo

INTERVENTIONS:
Other: SH-DS01 + Antibiotic Placebo — Participants will be instructed to take 2 capsules of SH-DS01 probiotic once daily (at lunch) from cycle day 1 to the day of ovulation/day of luteal progesterone initiation, followed by 2 capsules of SH-DS01 probiotic once daily (at lunch) and 1 capsule of placebo for antibiotic twice daily (at breakfast and dinner) from the day of ovulation/day of luteal progesterone initiation to the day of frozen embryo transfer.
  Arms: Probiotic + Antibiotic Placebo
Drug: SH-DS01 + Metronidazole — Participants will be instructed to take 2 capsules of SH-DS01 probiotic once daily (at lunch) from cycle day 1 to the day of ovulation/day of luteal progesterone initiation, followed by 2 capsules of SH-DS01 probiotic once daily (at lunch) and 1 capsule of 500mg metronidazole twice daily (at breakfast and dinner) from the day of ovulation/day of luteal progesterone initiation to the day of frozen embryo transfer.
  Arms: Probiotic + Antibiotic
Other: Probiotic Placebo + Antibiotic Placebo — Participants will be instructed to take 2 capsules of placebo for probiotic once daily (at lunch) from cycle day 1 to the day of ovulation/day of luteal progesterone initiation, followed by 2 capsules of placebo for probiotic once daily (at lunch) and 1 capsule of placebo for antibiotic twice daily (at breakfast and dinner) from the day of ovulation/day of luteal progesterone initiation to the day of frozen embryo transfer.
  Arms: Probiotic Placebo + Antibiotic Placebo

SUMMARY:
The study is designed as a proof of concept pilot study with 3 study arms to evaluate the safety and feasibility of the use of oral probiotics and/or antibiotics in women with unexplained infertility/endometriosis. Our secondary outcomes will assess In Vitro Fertilization outcomes, and changes in the uterine microbiota (bacteria), intestinal barrier integrity, and urinary metabolites in response to study interventions.

DETAILED DESCRIPTION:
Previous research has demonstrated that the uterine microbiota can impact fertility and embryo implantation. This information leads to the hypothesis that prophylactic antibiotic and/or probiotic treatment may improve reproductive outcomes in women with unexplained infertility/endometriosis who are seeking In Vitro Fertilization (IVF). No therapeutic protocols to improve these outcomes currently exist. However, there are safe and easily accessible medications and supplements that may be able to optimally modify the uterine microbiota. Herein we are proposing a proof of concept pilot study of the feasibility, safety and tolerability of administering oral probiotics, or oral probiotics in combination with antibiotics, to women seeking IVF.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged 18-40 at the time of egg retrieval
2. Generally in good health (at physician's discretion)
3. Diagnosed with Unexplained Infertility
4. Diagnosed with or suspected of having endometriosis (at ONE Fertility physician's discretion)
5. Normal uterine cavity as assessed by prior sonohysterogram
6. Planning to undergo Frozen Embryo Transfer with ≥1 frozen blastocyst ≥3BB (grade Gardner) to transfer
7. Able to understand, comply and consent to protocol requirements and instructions
8. Able to attend scheduled study visits and complete required investigations

Exclusion Criteria:

1. Any known endometrial pathologies other than endometriosis
2. Polycystic ovary syndrome
3. Ovulatory dysfunction
4. Male factor infertility (Total Motile Sperm Count <5M/mL)
5. Poorly controlled auto-immune disease and/or diabetes (at physician's discretion)
6. Is immune-compromised
7. Cockayne syndrome
8. Allergy to Metronidazole
9. Allergy to rice (bran and hull), pomegranate, Acacia gum, hypromellose, fermented gellan gum, chlorophyllin, or sunflower oil
10. Known intolerance of Lactobacillus and/or Bifidobacterium-containing probiotics
11. Antibiotic use in the past month
12. Use of any of the following:

    1. Oral probiotics
    2. Alcohol
    3. Anticoagulant therapies (Warfarin type)
    4. Drugs containing alcohol
    5. Busulfan
    6. Cyclosporin
    7. Disulfiram
    8. 5-Fluoruracil
    9. Lithium
    10. Phenytoin or Phenobarbital
    11. Vecuronium
    12. Proton pump inhibitors
    13. Histamine H2-receptor antagonists
13. Currently experiencing nausea, fever, vomiting, bloody diarrhea or severe abdominal pain

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Rate of study enrollment | Screening
  Evaluated by number of eligible participants consenting to enrollment in the study.
Rate of retention of study participants | Immediately after the intervention
  Evaluated by number of study participants who complete, drop out or withdraw from the study.
Proportion of participants adhering to study protocol | Immediately after the intervention
  Evaluated as the percentage of study participants reporting daily administration of study interventions throughout the intervention period.
Incidence of intervention-emergent adverse events | Immediately after the intervention
  Evaluated as the percentage of adverse events occurring in each intervention group.

SECONDARY OUTCOMES:
Difference in implantation rate | Endpoint of interventions to 4 weeks gestation (if applicable)
  Evaluated by number of people with a positive beta hCG 2 weeks following frozen embryo transfer (FET), between intervention groups.
Difference in clinical pregnancy rate | Endpoint of interventions to 6 weeks gestation (if applicable)
  Evaluated by number of people with a clinical pregnancy (gestational sac with fetal pole and cardiac activity seen on ultrasound at 6 weeks gestation), between intervention groups.
Difference in ongoing pregnancy rate | Endpoint of interventions to 12 weeks gestation (if applicable)
  Evaluated by number of people with an ongoing pregnancy (gestational sac with fetal pole and cardiac activity seen on ultrasound at 12 weeks gestation), between intervention groups.
Change in uterine microbiota composition | Baseline, immediately after interventions
  Evaluated by 16S rRNA sequencing of the uterine microbiota at baseline versus on the day of FET, and compared between experimental groups.
Change in serum LPS | Baseline, immediately after interventions
  Evaluated by changes in LPS-binding protein (LPS) at baseline versus on the day of FET, and compared between intervention groups.
Change in intestinal permeability | Baseline, immediately after interventions
  Evaluated by changes in untargeted peripheral blood metabolites at baseline versus on the day of FET, and compared between intervention groups.
Change in peripheral cytokines | Baseline, immediately after interventions
  Evaluated by changes in peripheral cytokines (TNF, IL-6, IL-8, IFNg - in pg/mL) at baseline versus on the day of FET, and compared between intervention groups.
Change in urinary metabolites | Baseline, immediately after interventions
  Evaluated by changes untargeted urinary metabolites at baseline versus on the day of FET, and compared between intervention groups. Nontargeted metabolic phenotyping of >100 urinary metabolites will be performed by multisegment injection capillary electrophoresis-mass spectrometry (MSI-CE-MS) as a high throughput platform to analyze metabolites. The fold change for each metabolite will be calculated between baseline vs. after interventions, and the fold changes will be compared between intervention groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn Wessels, PhD, Principal Investigator — McMaster University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eckert LO, Moore DE, Patton DL, Agnew KJ, Eschenbach DA. Relationship of vaginal bacteria and inflammation with conception and early pregnancy loss following in-vitro fertilization. Infect Dis Obstet Gynecol. 2003;11(1):11-7. doi: 10.1155/S1064744903000024. PMID 12839628
- [Background] Selman H, Mariani M, Barnocchi N, Mencacci A, Bistoni F, Arena S, Pizzasegale S, Brusco GF, Angelini A. Examination of bacterial contamination at the time of embryo transfer, and its impact on the IVF/pregnancy outcome. J Assist Reprod Genet. 2007 Sep;24(9):395-9. doi: 10.1007/s10815-007-9146-5. Epub 2007 Jul 17. PMID 17636439
- [Background] Moreno I, Codoner FM, Vilella F, Valbuena D, Martinez-Blanch JF, Jimenez-Almazan J, Alonso R, Alama P, Remohi J, Pellicer A, Ramon D, Simon C. Evidence that the endometrial microbiota has an effect on implantation success or failure. Am J Obstet Gynecol. 2016 Dec;215(6):684-703. doi: 10.1016/j.ajog.2016.09.075. Epub 2016 Oct 4. PMID 27717732
- [Background] Kyono K, Hashimoto T, Nagai Y, Sakuraba Y. Analysis of endometrial microbiota by 16S ribosomal RNA gene sequencing among infertile patients: a single-center pilot study. Reprod Med Biol. 2018 May 6;17(3):297-306. doi: 10.1002/rmb2.12105. eCollection 2018 Jul. PMID 30013432
- [Background] Fanchin R, Harmas A, Benaoudia F, Lundkvist U, Olivennes F, Frydman R. Microbial flora of the cervix assessed at the time of embryo transfer adversely affects in vitro fertilization outcome. Fertil Steril. 1998 Nov;70(5):866-70. doi: 10.1016/s0015-0282(98)00277-5. PMID 9806568
- [Background] Egbase PE, Udo EE, Al-Sharhan M, Grudzinskas JG. Prophylactic antibiotics and endocervical microbial inoculation of the endometrium at embryo transfer. Lancet. 1999 Aug 21;354(9179):651-2. doi: 10.1016/s0140-6736(99)02415-0. PMID 10466674
- [Background] Moore DE, Soules MR, Klein NA, Fujimoto VY, Agnew KJ, Eschenbach DA. Bacteria in the transfer catheter tip influence the live-birth rate after in vitro fertilization. Fertil Steril. 2000 Dec;74(6):1118-24. doi: 10.1016/s0015-0282(00)01624-1. PMID 11119737
- [Background] Brook N, Khalaf Y, Coomarasamy A, Edgeworth J, Braude P. A randomized controlled trial of prophylactic antibiotics (co-amoxiclav) prior to embryo transfer. Hum Reprod. 2006 Nov;21(11):2911-5. doi: 10.1093/humrep/del263. Epub 2006 Jul 10. PMID 16832124